CLINICAL TRIAL: NCT00127855
Title: A Phase II, Open (Partially Double-blind), Randomised, Controlled, Multicentre, Primary Vaccination Study to Evaluate the Immunogenicity (Including Immune Memory), Reactogenicity and Safety of Three Different Formulations of the GSK Biologicals' Combined Haemophilus Influenzae Type B-meningococcal Serogroups CY Conjugate Vaccine Given Concomitantly With Infanrix® Penta and Prevenar®, Versus ActHIB® and Meningitec® Given Concomitantly With Infanrix® Penta and Versus ActHIB® Given Concomitantly With Infanrix® Penta and Prevenar® in Infants According to a 2-4-6 Month Schedule.
Brief Title: Dose Ranging Study of Combined Haemophilus Influenzae Type B-Meningococcal Serogroups CY (Hib-MenCY-TT) Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 792014/001; 792014/002 (Other: GSK)
Record Dates: First submitted 2005-08-08; First posted 2005-08-09 (Estimated); Results first posted 2012-07-23 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2016-10

CONDITIONS: Haemophilus Influenzae Type b; Neisseria Meningitidis
Keywords: Invasive bacterial disease caused by Hib; Neisseria meningitidis serogroups C & Y
MeSH Terms: conditions — Haemophilus Infections | interventions — Hib-MenCY-TT vaccine; Haemophilus influenza type b polysaccharide vaccine-tetanus toxin conjugate; DTPa-HBV-IPV combined vaccine; Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (5):
- MenHibrix Formulation 1 Group (Experimental): Subjects were primed with MenHibrix formulation 1 co-administered with Infanrix Penta and Prevenar according to a 2-4-6 months of age schedule, and received a polysaccharide challenge dose (1/5th dose of MenACWY polysaccharide vaccine co-administered with 10 µg dose of plain PRP) at 12 months of age.
  Interventions: Biological: Hib-MenCY-TT vaccine (MenHibrix); Biological: Infanrix® Penta; Biological: Prevenar®; Biological: Mencevax® ACWY; Biological: PRP (Polyribosyl Ribitol Phosphate)
- MenHibrix Formulation 2 Group (Experimental): Subjects were primed with MenHibrix formulation 2 co-administered with Infanrix Penta and Prevenar according to a 2-4-6 months of age schedule, and received a polysaccharide challenge dose (1/5th dose of MenACWY polysaccharide vaccine co-administered with 10 µg dose of plain PRP) at 12 months of age.
  Interventions: Biological: Hib-MenCY-TT vaccine (MenHibrix); Biological: Infanrix® Penta; Biological: Prevenar®; Biological: Mencevax® ACWY; Biological: PRP (Polyribosyl Ribitol Phosphate)
- MenHibrix Formulation 3 Group (Experimental): Subjects were primed with MenHibrix formulation 3 co-administered with Infanrix Penta and Prevenar according to a 2-4-6 months of age schedule, and received a polysaccharide challenge dose (1/5th dose of MenACWY polysaccharide vaccine co-administered with 10 µg dose of plain PRP) at 12 months of age.
  Interventions: Biological: Hib-MenCY-TT vaccine (MenHibrix); Biological: Infanrix® Penta; Biological: Prevenar®; Biological: Mencevax® ACWY; Biological: PRP (Polyribosyl Ribitol Phosphate)
- Menjugate Group (Active Comparator): Subjects were primed with Menjugate co-administered with Infanrix Penta and ActiHIB according to a 2-4-6 months of age schedule, and received a polysaccharide challenge dose (1/5th dose of MenACWY polysaccharide vaccine co-administered with 10 µg dose of plain PRP) at 12 months of age.
  Interventions: Biological: Meningitec®; Biological: ActHIB®; Biological: Infanrix® Penta; Biological: Mencevax® ACWY; Biological: PRP (Polyribosyl Ribitol Phosphate)
- ActHIB Group (Active Comparator): Subjects were primed with ActHIB co-administered with Infanrix Penta and Prevenar according to a 2-4-6 months of age schedule, and received a polysaccharide challenge dose (1/5th dose of MenACWY polysaccharide vaccine co-administered with 10 µg dose of plain PRP) at 12 months of age.
  Interventions: Biological: ActHIB®; Biological: Infanrix® Penta; Biological: Prevenar®; Biological: Mencevax® ACWY; Biological: PRP (Polyribosyl Ribitol Phosphate)

INTERVENTIONS:
Biological: Hib-MenCY-TT vaccine (MenHibrix) — Three doses were administered intramuscularly (IM) in left thigh at Months 0,2 and 4 respectively
  Arms: MenHibrix Formulation 1 Group; MenHibrix Formulation 2 Group; MenHibrix Formulation 3 Group
Biological: Meningitec® — Three doses were administered IM in right lower thigh at Months 0,2 and 4.
  Arms: Menjugate Group
Biological: ActHIB® — Three doses were administered IM in left thigh at Months 0,2 and 4.
  Arms: ActHIB Group; Menjugate Group
Biological: Infanrix® Penta — Three doses were administered IM in right upper thigh at Months 0,2 and 4 respectively.
  Other Names: DTPa-HBV-IPV vaccine
Biological: Prevenar® — Three doses were administered IM in right lower thigh at Months 0,2 and 4 respectively.
  Arms: ActHIB Group; MenHibrix Formulation 1 Group; MenHibrix Formulation 2 Group; MenHibrix Formulation 3 Group
Biological: Mencevax® ACWY — One fifth of one dose was administered IM in deltoid region of right arm at Month 10 as booster.
Biological: PRP (Polyribosyl Ribitol Phosphate) — One dose was administered IM in deltoid region of left arm at Month 10 as booster.

SUMMARY:
This study evaluated the safety and immunogenicity of 3 formulations of Hib-MenCY-TT vaccine compared to 2 control groups receiving licensed meningococcal serogroup C conjugate vaccine and/or licensed Hib conjugate vaccine administered at 2, 4, and 6 months of age. Antibody persistence and immune responses to polysaccharide vaccine boosters were additionally assessed at 11 to 14 months of age.

ELIGIBILITY:
Inclusion criteria:

* A male or female between, and including, 6 and 12 weeks (42-90 days) of age at the time of the first vaccination.
* Written informed consent obtained from the parent or guardian of the subject.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.
* Vaccinated against hepatitis B at birth.
* Born after a gestation period of 36 - 42 weeks.

Exclusion criteria:

* Use of any investigational or non-registered drug or vaccine other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs since birth
* Any chronic drug therapy to be continued during the study period.
* Planned administration/ administration of a vaccine not foreseen by the study protocol within one month of the first dose of vaccine(s).
* Previous vaccination against diphtheria, tetanus, pertussis, polio, N. meningitidis of serogroups C and Y, Haemophilus influenzae type b or Streptococcus pneumoniae.
* History of or known exposure to diphtheria, tetanus, pertussis, polio, or invasive diseases due to N. meningitidis of serogroups C and Y, Haemophilus influenzae type b or Streptococcus pneumoniae.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.
* A family history of congenital or hereditary immunodeficiency.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines.
* Major congenital defects or serious chronic illness.
* History of any neurologic disorders or seizures.
* Acute disease at the time of enrolment.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 409 (Actual)
Dates: Start 2003-03-01; Primary Completion 2004-02-01 (Actual); Study Completion 2004-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- Australia (3):
  - GSK Investigational Site, North Adelaide, South Australia
  - GSK Investigational Site, Carlton, Victoria
  - GSK Investigational Site, Subiaco, Western Australia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Bryant KA, Marshall GS. Haemophilus influenzae type b-Neisseria meningitidis serogroups C and Y tetanus toxoid conjugate vaccine for infants and toddlers. Expert Rev Vaccines. 2011 Jul;10(7):941-50. doi: 10.1586/erv.11.90. PMID 21806393
- [Background] Nolan T, Lambert S, Roberton D, Marshall H, Richmond P, Streeton C, Poolman J, Boutriau D. A novel combined Haemophilus influenzae type b-Neisseria meningitidis serogroups C and Y-tetanus-toxoid conjugate vaccine is immunogenic and induces immune memory when co-administered with DTPa-HBV-IPV and conjugate pneumococcal vaccines in infants. Vaccine. 2007 Dec 12;25(51):8487-99. doi: 10.1016/j.vaccine.2007.10.013. Epub 2007 Oct 25. PMID 17996996
- [Background] T Nolan et al. A novel Haemophilus influenzae type b - meningococcal serogroups C and Y conjugate (Hib-MenCY-TT) vaccine induces persistent immune responses and immune memory. Abstract presented at Pediatric Academic Societies' (PAS) Annual meeting. San Francisco, California, US, 29 April to 2 May 2006.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 792014/001 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 792014/001 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 792014/001 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 792014/001 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 792014/001 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 409 subjects enrolled, two subjects were determined to be ineligible for enrolment and were actually never vaccinated. Not all subjects that started the primary vaccination course returned for the polysaccharide challenge dose administration.
Period: Primary Vaccination Course
Arm/Group | MenHibrix Formulation 1 Group | MenHibrix Formulation 2 Group | MenHibrix Formulation 3 Group | Menjugate Group | ActHIB Group
Started | 82 | 82 | 80 | 81 | 82
Completed | 80 | 81 | 78 | 81 | 78
Not Completed | 2 | 1 | 2 | 0 | 4
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 1 | 1 | 0 | 2
Not completed — Other | 0 | 0 | 0 | 0 | 1
Period: Polysaccharide Challenge Dose
Arm/Group | MenHibrix Formulation 1 Group | MenHibrix Formulation 2 Group | MenHibrix Formulation 3 Group | Menjugate Group | ActHIB Group
Started | 80 | 79 | 77 | 81 | 77
Completed | 80 | 79 | 77 | 81 | 77
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MenHibrix Formulation 1 Group | MenHibrix Formulation 2 Group | MenHibrix Formulation 3 Group | Menjugate Group | ActHIB Group | Total
Number analyzed (Participants) | 82 | 82 | 80 | 81 | 82 | 407
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 8.1 (1.39) | 8.3 (1.46) | 8.2 (1.65) | 8.0 (1.65) | 8.1 (1.43) | 8.1 (1.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 45 | 41 | 43 | 37 | 204
  Male | 44 | 37 | 39 | 38 | 45 | 203

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Anti-polyribosyl Ribitol Phosphate (Anti-PRP) Antibody Concentrations Greater Than or Equal to 1 Milligram Per Milliliter
Description: The cut-off concentration assessed was 1 milligram per milliliter (mg/mL).
Time Frame: One month after primary vaccination (Month 5)
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, including all evaluable subjects for whom assay results were available for antibodies against at least one study vaccine antigen component, for at least one blood sample during the primary vaccination course.
Measure: Number; unit: Subjects
Arm/Group | MenHibrix Formulation 1 Group | MenHibrix Formulation 2 Group | MenHibrix Formulation 3 Group | Menjugate Group | ActHIB Group
Number analyzed (Participants) | 74 | 76 | 70 | 74 | 74
Subjects | 72 | 75 | 65 | 66 | 70

2. Primary Outcome: Number of Subjects With Serum Bactericidal Activity Using Baby Rabbit Complement (rSBA)- Neisseria Meningitidis Serogroup C (MenC) Titers Greater Than or Equal to 1:8
Description: The cut-off titer assessed was a dilution of 1:8. Titers were expressed as the reciprocal of the dilution resulting in 50 percent inhibition.
Time Frame: One month after primary vaccination (Month 5)
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | MenHibrix Formulation 1 Group | MenHibrix Formulation 2 Group | MenHibrix Formulation 3 Group | Menjugate Group | ActHIB Group
Number analyzed (Participants) | 69 | 76 | 72 | 74 | 76
Subjects | 69 | 76 | 72 | 74 | 1

3. Primary Outcome: Number of Subjects With Serum Bactericidal Activity Using Baby Rabbit Complement (rSBA)- Neisseria Meningitidis Serogroup Y (MenY) Titers Greater Than or Equal to 1:8
Description: as for outcome 2
Time Frame: One month after primary vaccination (Month 5)
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | MenHibrix Formulation 1 Group | MenHibrix Formulation 2 Group | MenHibrix Formulation 3 Group | Menjugate Group | ActHIB Group
Number analyzed (Participants) | 67 | 68 | 69 | 68 | 74
Subjects | 66 | 68 | 68 | 10 | 12

4. Secondary Outcome: Number of Subjects With Serum Bactericidal Activity Using Baby Rabbit Complement (rSBA)- Neisseria Meningitidis Serogroup C (MenC) Titers Greater Than or Equal to 1:8
Description: as for outcome 2
Time Frame: Prior to vaccination (Day 0), before administration of the polysaccharide challenge dose (Month 10) and one month after administration of the polysaccharide challenge dose (Month 11)
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity for Day 0 data and on the Booster ATP cohort for immunogenicity for the Month 10/Month 11 data.
Measure: Number; unit: Subjects
Arm/Group | MenHibrix Formulation 1 Group | MenHibrix Formulation 2 Group | MenHibrix Formulation 3 Group | Menjugate Group | ActHIB Group
Number analyzed (Participants) | 69 | 73 | 73 | 79 | 70
Subjects
  Day 0 (N= 68; 66; 63; 66; 70) | 2 | 6 | 2 | 3 | 1
  Month 10 (N= 69; 71; 73; 74; 68) | 67 | 70 | 70 | 67 | 6
  Month 11 (N= 69; 73; 71; 79; 66) | 69 | 73 | 71 | 77 | 18

5. Secondary Outcome: Serum Bactericidal Activity Using Baby Rabbit Complement (rSBA)- Neisseria Meningitidis Serogroup C (MenC) Titers
Description: Titers were presented as geometric mean titers (GMTs) expressed as the reciprocal of the dilution resulting in 50 percent inhibition.
Time Frame: Prior to vaccination (Day 0), one month after the 3-dose primary vaccination course (Month 5), before administration of the polysaccharide challenge dose (Month 10) and one month after administration of the polysaccharide challenge dose (Month 11)
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity for Day 0/Month5 data and on the Booster ATP cohort for immunogenicity for the Month 10/Month 11 data.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | MenHibrix Formulation 1 Group | MenHibrix Formulation 2 Group | MenHibrix Formulation 3 Group | Menjugate Group | ActHIB Group
Number analyzed (Participants) | 69 | 76 | 73 | 79 | 76
Titer
  Day 0 (N= 68; 66; 63; 66; 70) | 4.3 [3.9 to 4.7] | 5.2 [4.1 to 6.6] | 4.2 [3.9 to 4.6] | 4.2 [4.0 to 4.5] | 4.1 [3.9 to 4.4]
  Month 5 (N= 69; 76; 72; 74; 76) | 1293.1 [1027.7 to 1627.1] | 1065.6 [858.8 to 1322.3] | 968.4 [770.8 to 1216.6] | 1931.9 [1541.2 to 2421.6] | 4.2 [3.8 to 4.5]
  Month 10 (N= 69; 71; 73; 74; 68) | 260.5 [190.7 to 355.8] | 214.2 [163.5 to 280.7] | 199.8 [143.8 to 277.6] | 170.8 [113.2 to 257.7] | 4.9 [4.2 to 5.7]
  Month 11 (N= 69; 73; 71; 79; 66) | 1985.5 [1542.6 to 2555.8] | 919.5 [692.3 to 1221.2] | 1530.4 [1119.6 to 2091.8] | 774.8 [536.7 to 1118.5] | 9.0 [6.4 to 12.8]

6. Secondary Outcome: Number of Subjects With rSBA-MenY Titers Greater Than or Equal to 1:8
Description: as for outcome 2
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Number; unit: Subjects
Arm/Group | MenHibrix Formulation 1 Group | MenHibrix Formulation 2 Group | MenHibrix Formulation 3 Group | Menjugate Group | ActHIB Group
Number analyzed (Participants) | 69 | 71 | 70 | 77 | 71
Subjects
  Day 0 (N= 68; 65; 58; 63; 66) | 4 | 7 | 5 | 9 | 4
  Month 10 (N= 69; 69; 70; 71; 68) | 61 | 55 | 60 | 17 | 22
  Month 11 (N= 68; 71; 70; 77; 71) | 68 | 71 | 69 | 32 | 38

7. Secondary Outcome: Serum Bactericidal Activity Using Baby Rabbit Complement (rSBA)- Neisseria Meningitidis Serogroup Y (MenY) Titers
Description: as for outcome 5
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | MenHibrix Formulation 1 Group | MenHibrix Formulation 2 Group | MenHibrix Formulation 3 Group | Menjugate Group | ActHIB Group
Number analyzed (Participants) | 69 | 71 | 70 | 77 | 74
Titer
  Day 0 (N= 68; 65; 58; 63; 66) | 4.6 [4.0 to 5.4] | 5.6 [4.3 to 7.2] | 5.1 [4.1 to 6.3] | 6.3 [4.7 to 8.4] | 4.9 [4.0 to 5.9]
  Month 5 (N= 67; 68; 69; 68; 74) | 843.5 [640.1 to 1111.7] | 1020.0 [790.0 to 1316.8] | 741.8 [538.0 to 1022.9] | 6.9 [5.0 to 9.5] | 7.3 [5.2 to 10.1]
  Month 10 (N= 69; 69; 70; 71; 68) | 114.5 [78.6 to 167.0] | 139.6 [86.8 to 224.7] | 129.9 [87.1 to 193.7] | 10.0 [6.7 to 15.0] | 13.4 [8.6 to 20.9]
  Month 11 (N= 68; 71; 70; 77; 71) | 1838.0 [1427.9 to 2366.0] | 1539.8 [1165.4 to 2034.5] | 1653.8 [1202.5 to 2274.4] | 18.8 [12.1 to 29.4] | 32.0 [19.7 to 52.0]

8. Secondary Outcome: Number of Subjects With Anti-polysaccharide C (PSC) Antibody Concentration Greater Than or Equal to 30 Micrograms Per Milliliter (µg/mL)
Description: The cut-off concentration assessed was 30 micrograms per milliliter (µg/mL).
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Number; unit: Subjects
Arm/Group | MenHibrix Formulation 1 Group | MenHibrix Formulation 2 Group | MenHibrix Formulation 3 Group | Menjugate Group | ActHIB Group
Number analyzed (Participants) | 71 | 70 | 71 | 76 | 71
Subjects
  Day 0 (N= 54; 54; 49; 56; 56) | 5 | 5 | 6 | 5 | 4
  Month 5 (N= 63; 65; 61; 62; 63) | 63 | 65 | 61 | 62 | 1
  Month 10 (N= 63; 68; 61; 74; 67) | 63 | 68 | 61 | 74 | 1
  Month 11 (N= 71; 70; 71; 76; 71) | 71 | 70 | 71 | 76 | 69

9. Secondary Outcome: Anti-polysaccharide C (PSC) Antibody Concentration
Description: Titers are presented as Geometric Mean Titers (GMTs) expressed as micrograms per milliliter (µg/mL).
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: microgram per milliliter (µg/mL)
Arm/Group | MenHibrix Formulation 1 Group | MenHibrix Formulation 2 Group | MenHibrix Formulation 3 Group | Menjugate Group | ActHIB Group
Number analyzed (Participants) | 71 | 70 | 71 | 76 | 71
microgram per milliliter (µg/mL)
  Day 0 (N= 54; 54; 49; 56; 56) | 0.17 [0.15 to 0.20] | 0.17 [0.15 to 0.18] | 0.17 [0.15 to 0.19] | 0.17 [0.15 to 0.20] | 0.17 [0.15 to 0.19]
  Month 5 (N= 63; 65; 61; 62; 63) | 12.02 [9.90 to 14.59] | 12.09 [10.59 to 13.81] | 9.95 [8.34 to 11.87] | 15.36 [12.67 to 18.62] | 0.15 [0.15 to 0.16]
  Month 10 (N= 63; 68; 61; 74; 67) | 3.11 [2.52 to 3.85] | 3.10 [2.64 to 3.64] | 2.74 [2.29 to 3.27] | 2.87 [2.23 to 3.71] | 0.15 [0.15 to 0.16]
  Month 11 (N= 71; 70; 71; 76; 71) | 11.47 [9.25 to 14.22] | 7.94 [6.42 to 9.81] | 10.96 [8.63 to 13.91] | 7.56 [6.17 to 9.26] | 1.49 [1.23 to 1.81]

10. Secondary Outcome: Number of Subjects With Anti-polysaccharide Y (PSY) Antibody Concentration Greater Than or Equal to 30 Micrograms Per Milliliter (µg/mL)
Description: The cut-off concentration assessed was 30 micrograms per milliliter (µg/mL).
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Number; unit: Subjects
Arm/Group | MenHibrix Formulation 1 Group | MenHibrix Formulation 2 Group | MenHibrix Formulation 3 Group | Menjugate Group | ActHIB Group
Number analyzed (Participants) | 70 | 71 | 72 | 77 | 71
Subjects
  Day 0 (N= 51; 51; 47; 56; 54) | 3 | 4 | 3 | 7 | 7
  Month 5 (N= 67; 70; 72; 66; 69) | 67 | 70 | 72 | 2 | 0
  Month 10 (N= 70; 69; 71; 76; 67) | 70 | 69 | 70 | 0 | 1
  Month 11 (N= 69; 71; 71; 77; 71) | 69 | 71 | 71 | 70 | 64

11. Secondary Outcome: Anti-polysaccharide Y (PSY) Antibody Concentration
Description: Titers are presented as Geometric Mean Titers (GMTs) expressed as micrograms per milliliter (µg/mL).
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Microgram per milliliter (µg/mL)
Arm/Group | MenHibrix Formulation 1 Group | MenHibrix Formulation 2 Group | MenHibrix Formulation 3 Group | Menjugate Group | ActHIB Group
Number analyzed (Participants) | 70 | 71 | 72 | 77 | 71
Microgram per milliliter (µg/mL)
  Day 0 (N= 51; 51; 47; 56; 54) | 0.17 [0.15 to 0.19] | 0.18 [0.15 to 0.23] | 0.17 [0.15 to 0.19] | 0.20 [0.16 to 0.26] | 0.19 [0.16 to 0.23]
  Month 5 (N= 67; 70; 72; 66; 69) | 19.22 [15.42 to 23.95] | 19.09 [15.44 to 23.59] | 15.83 [12.64 to 19.82] | 0.16 [0.15 to 0.17] | 0.15 [0.15 to 0.15]
  Month 10 (N= 70; 69; 71; 76; 67) | 5.26 [4.20 to 6.60] | 5.20 [4.17 to 6.49] | 4.10 [3.22 to 5.23] | 0.15 [0.15 to 0.15] | 0.15 [0.15 to 0.16]
  Month 11 (N= 69; 71; 71; 77; 71) | 47.95 [39.80 to 57.77] | 37.15 [29.16 to 47.32] | 51.12 [38.71 to 67.52] | 1.37 [1.05 to 1.79] | 1.33 [1.02 to 1.72]

12. Secondary Outcome: Number of Subjects With Anti-PRP Antibody Concentration Greater Than or Equal to Pre-defined Cut-off Values
Description: The cut-off concentrations assessed were 0.15 micrograms per milliliter (µg/mL) and 1 µg/mL.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Number; unit: Subjects
Arm/Group | MenHibrix Formulation 1 Group | MenHibrix Formulation 2 Group | MenHibrix Formulation 3 Group | Menjugate Group | ActHIB Group
Number analyzed (Participants) | 74 | 76 | 73 | 79 | 74
Subjects
  Day 0 ≥ 0.15 µg/mL (N= 68; 70; 67; 67; 73) | 29 | 37 | 41 | 32 | 37
  Month 5 ≥ 0.15 µg/mL (N= 74; 76; 70; 74; 74) | 74 | 76 | 70 | 73 | 74
  Month 10 ≥ 0.15 µg/mL (N= 70; 72; 73; 76; 70) | 70 | 71 | 72 | 71 | 68
  Month 11 ≥ 0.15 µg/mL (N= 68; 73; 71; 79; 72) | 68 | 72 | 71 | 78 | 71
  Day 0 ≥ 1 µg/mL (N= 68; 70; 67; 67; 73) | 7 | 10 | 6 | 6 | 8
  Month 5 ≥ 1 µg/mL (N= 74; 76; 70; 74; 74) | 72 | 75 | 65 | 66 | 70
  Month 10 ≥ 1 µg/mL (N= 70; 72; 73; 76; 70) | 46 | 42 | 36 | 39 | 41
  Month 11 ≥ 1 µg/mL (N= 68; 73; 71; 79; 72) | 67 | 69 | 65 | 57 | 58

13. Secondary Outcome: Anti-PRP Antibody Concentration
Description: Concentrations are presented as GMCs and expressed as µg/mL.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Microgram per milliliter (µg/mL)
Arm/Group | MenHibrix Formulation 1 Group | MenHibrix Formulation 2 Group | MenHibrix Formulation 3 Group | Menjugate Group | ActHIB Group
Number analyzed (Participants) | 74 | 76 | 73 | 79 | 74
Microgram per milliliter (µg/mL)
  Day 0 (N= 68; 70; 67; 67; 73) | 0.152 [0.120 to 0.194] | 0.224 [0.164 to 0.305] | 0.214 [0.166 to 0.276] | 0.172 [0.132 to 0.223] | 0.201 [0.153 to 0.265]
  Month 5 (N= 74; 76; 70; 74; 74) | 6.441 [5.315 to 7.805] | 7.324 [5.877 to 9.127] | 5.577 [4.375 to 7.110] | 4.465 [3.399 to 5.865] | 5.714 [4.538 to 7.195]
  Month 10 (N= 70; 72; 73; 76; 70) | 1.386 [1.134 to 1.693] | 1.383 [1.092 to 1.751] | 1.148 [0.914 to 1.441] | 0.949 [0.728 to 1.238] | 1.141 [0.868 to 1.501]
  Month 11 (N= 68; 73; 71; 79; 72) | 8.653 [6.701 to 11.173] | 6.750 [5.002 to 9.107] | 5.112 [3.878 to 6.739] | 2.512 [1.837 to 3.435] | 3.283 [2.380 to 4.529]

14. Secondary Outcome: Number of Subjects Seroprotected for Anti-diphtheria Antibodies
Description: Seroprotection is defined as anti-diphtheria toxoid antibody concentration greater than or equal to 0.1 International Units per Milliliter (IU/mL).
Time Frame: Prior to vaccination (Day 0), one month after the 3-dose primary vaccination course (Month 5) and before administration of the polysaccharide challenge dose (Month 10)
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity for Day 0/Month5 data and on the Booster ATP cohort for safety, including all vaccinated subjects who had not received a vaccine not specified or forbidden in the protocol, for the Month 10 data.
Measure: Number; unit: Subjects
Arm/Group | MenHibrix Formulation 1 Group | MenHibrix Formulation 2 Group | MenHibrix Formulation 3 Group | Menjugate Group | ActHIB Group
Number analyzed (Participants) | 78 | 78 | 75 | 80 | 76
Subjects
  Day 0 (N= 68; 70; 65; 69; 74) | 26 | 28 | 28 | 26 | 29
  Month 5 (N= 74; 76; 74; 77; 76) | 74 | 76 | 74 | 77 | 76
  Month 10 (N= 78; 78; 75; 80; 75) | 76 | 75 | 72 | 74 | 75

15. Secondary Outcome: Anti-diphtheria Antibody Concentrations
Description: Concentrations are presented as GMCs and expressed as International Units per Milliliter (IU/mL).
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: International Units per Milliliter
Arm/Group | MenHibrix Formulation 1 Group | MenHibrix Formulation 2 Group | MenHibrix Formulation 3 Group | Menjugate Group | ActHIB Group
Number analyzed (Participants) | 78 | 78 | 75 | 80 | 76
International Units per Milliliter
  Day 0 (N= 68; 70; 65; 69; 74) | 0.090 [0.074 to 0.110] | 0.098 [0.077 to 0.123] | 0.101 [0.080 to 0.127] | 0.090 [0.074 to 0.110] | 0.093 [0.074 to 0.117]
  Month 5 (N= 74; 76; 74; 77; 76) | 1.721 [1.480 to 2.003] | 1.797 [1.508 to 2.141] | 2.000 [1.706 to 2.346] | 1.845 [1.598 to 2.130] | 1.970 [1.760 to 2.206]
  Month 10 (N= 78; 78; 75; 80; 75) | 0.513 [0.423 to 0.622] | 0.505 [0.410 to 0.621] | 0.519 [0.423 to 0.638] | 0.405 [0.330 to 0.497] | 0.543 [0.467 to 0.631]

16. Secondary Outcome: Number of Subjects Seroprotected for Anti-tetanus Antibodies
Description: Seroprotection is defined as anti-tetanus toxoid antibody concentration greater than or equal to 0.1 International Units per Milliliter (IU/mL).
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Number; unit: Subjects
Arm/Group | MenHibrix Formulation 1 Group | MenHibrix Formulation 2 Group | MenHibrix Formulation 3 Group | Menjugate Group | ActHIB Group
Number analyzed (Participants) | 78 | 78 | 75 | 80 | 76
Subjects
  Day 0 (N= 62; 64; 60; 60; 68) | 54 | 58 | 57 | 57 | 62
  Month 5 (N= 74; 76; 74; 77; 76) | 74 | 76 | 74 | 77 | 76
  Month 10 (N= 78; 78; 75; 80; 75) | 78 | 78 | 74 | 78 | 75

17. Secondary Outcome: Anti-tetanus Antibody Concentrations
Description: Concentrations are presented as GMCs and expressed as International Units per Milliliter (IU/mL).
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: International Units per Milliliter
Arm/Group | MenHibrix Formulation 1 Group | MenHibrix Formulation 2 Group | MenHibrix Formulation 3 Group | Menjugate Group | ActHIB Group
Number analyzed (Participants) | 78 | 78 | 75 | 80 | 76
International Units per Milliliter
  Day 0 (N= 62; 64; 60; 60; 68) | 0.460 [0.343 to 0.617] | 0.470 [0.364 to 0.608] | 0.501 [0.386 to 0.651] | 0.562 [0.435 to 0.727] | 0.533 [0.403 to 0.705]
  Month 5 (N= 74; 76; 74; 77; 76) | 3.301 [2.909 to 3.747] | 3.816 [3.340 to 4.360] | 3.366 [2.974 to 3.810] | 1.877 [1.603 to 2.197] | 2.033 [1.773 to 2.330]
  Month 10 (N= 78; 78; 75; 80; 75) | 1.114 [0.967 to 1.283] | 1.307 [1.119 to 1.528] | 1.062 [0.905 to 1.246] | 0.603 [0.500 to 0.728] | 0.756 [0.633 to 0.902]

18. Secondary Outcome: Number of Subjects Seroseropositive for Anti-filamentus Haemagglutinin (FHA) Antibodies
Description: Seropositivity is defined as anti-FHA antibody concentration greater than or equal to 5 Enzyme-Linked Immunosorbent Assay (ELISA) Units per Milliliter (EL.U/mL).
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Number; unit: Subjects
Arm/Group | MenHibrix Formulation 1 Group | MenHibrix Formulation 2 Group | MenHibrix Formulation 3 Group | Menjugate Group | ActHIB Group
Number analyzed (Participants) | 78 | 78 | 75 | 79 | 76
Subjects
  Day 0 (N= 64; 69; 65; 67; 70) | 34 | 28 | 38 | 44 | 31
  Month 5 (N= 74; 76; 74; 77; 76) | 74 | 76 | 74 | 77 | 76
  Month 10 (N= 78; 78; 75; 79; 75) | 77 | 77 | 72 | 79 | 75

19. Secondary Outcome: Anti- FHA Antibody Concentrations
Description: Concentrations are presented as GMCs and expressed as Enzyme-Linked Immunosorbent Assay (ELISA) Units per Milliliter (EL.U/mL).
Time Frame: as for outcome 14
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity for Day 0/Month5 data and on the Booster ATP cohort for immunogenicity for the Month 10 data.
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA Units per Milliliter (EL.U/mL)
Arm/Group | MenHibrix Formulation 1 Group | MenHibrix Formulation 2 Group | MenHibrix Formulation 3 Group | Menjugate Group | ActHIB Group
Number analyzed (Participants) | 77 | 77 | 74 | 79 | 76
ELISA Units per Milliliter (EL.U/mL)
  Day 0 (N= 64; 69; 65; 67; 70) | 5.1 [4.2 to 6.2] | 4.6 [3.7 to 5.7] | 5.8 [4.8 to 7.1] | 7.4 [5.8 to 9.5] | 4.8 [3.9 to 5.9]
  Month 5 (N= 74; 76; 74; 77; 76) | 137.2 [116.4 to 161.7] | 141.5 [122.1 to 163.9] | 136.2 [118.0 to 157.2] | 132.1 [114.1 to 153.0] | 146.7 [124.8 to 172.4]
  Month 10 (N= 78; 78; 75; 79; 75) | 49.4 [40.6 to 60.0] | 50.9 [41.4 to 62.6] | 44.3 [35.7 to 55.0] | 39.9 [33.9 to 47.0] | 50.2 [41.6 to 60.6]

20. Secondary Outcome: Number of Subjects Seroseropositive for Anti-pertactin (PRN) Antibodies
Description: Seropositivity is defined as anti-PRN antibody concentration greater than or equal to 5 Enzyme-Linked Immunosorbent Assay (ELISA) Units per Milliliter (EL.U/mL).
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Number; unit: Subjects
Arm/Group | MenHibrix Formulation 1 Group | MenHibrix Formulation 2 Group | MenHibrix Formulation 3 Group | Menjugate Group | ActHIB Group
Number analyzed (Participants) | 78 | 78 | 75 | 80 | 76
Subjects
  Day 0 (N= 67; 63; 67; 68; 71) | 20 | 26 | 25 | 30 | 26
  Month 5 (N= 74; 76; 74; 77; 76) | 74 | 76 | 74 | 76 | 76
  Month 10 (N= 78; 78; 75; 80; 75) | 76 | 75 | 71 | 73 | 74

21. Secondary Outcome: Anti-PRN Antibody Concentrations
Description: as for outcome 19
Time Frame: as for outcome 14
Population: as for outcome 19
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA Units per Milliliter (EL.U/mL)
Arm/Group | MenHibrix Formulation 1 Group | MenHibrix Formulation 2 Group | MenHibrix Formulation 3 Group | Menjugate Group | ActHIB Group
Number analyzed (Participants) | 78 | 78 | 75 | 80 | 76
ELISA Units per Milliliter (EL.U/mL)
  Day 0 (N= 67; 63; 67; 68; 71) | 3.9 [3.2 to 4.7] | 4.7 [3.7 to 5.8] | 4.6 [3.7 to 5.7] | 5.3 [4.1 to 6.8] | 4.4 [3.6 to 5.4]
  Month 5 (N= 74; 76; 74; 77; 76) | 128.3 [107.4 to 153.1] | 120.7 [98.6 to 147.7] | 106.2 [89.3 to 126.3] | 112.9 [91.6 to 139.1] | 137.8 [118.2 to 160.7]
  Month 10 (N= 78; 78; 75; 80; 75) | 36.2 [29.5 to 44.3] | 31.8 [25.2 to 40.0] | 27.3 [22.1 to 33.8] | 27.2 [21.5 to 34.4] | 35.8 [29.7 to 43.1]

22. Secondary Outcome: Number of Subjects Seroseropositive for Anti-pertussis Toxoid (PT) Antibodies
Description: Seropositivity is defined as anti-PT antibody concentration greater than or equal to 5 Enzyme-Linked Immunosorbent Assay (ELISA) Units per Milliliter (EL.U/mL).
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Number; unit: Subjects
Arm/Group | MenHibrix Formulation 1 Group | MenHibrix Formulation 2 Group | MenHibrix Formulation 3 Group | Menjugate Group | ActHIB Group
Number analyzed (Participants) | 77 | 76 | 74 | 78 | 76
Subjects
  Day 0 (N= 65; 66; 65; 63; 74) | 5 | 6 | 5 | 11 | 3
  Month 5 (N= 74; 76; 74; 77; 76) | 74 | 76 | 74 | 77 | 76
  Month 10 (N= 77; 76; 73; 78; 75) | 71 | 66 | 62 | 61 | 63

23. Secondary Outcome: Anti- PT Antibody Concentrations
Description: as for outcome 19
Time Frame: as for outcome 14
Population: as for outcome 19
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA Units per Milliliter (EL.U/mL)
Arm/Group | MenHibrix Formulation 1 Group | MenHibrix Formulation 2 Group | MenHibrix Formulation 3 Group | Menjugate Group | ActHIB Group
Number analyzed (Participants) | 77 | 76 | 74 | 78 | 76
ELISA Units per Milliliter (EL.U/mL)
  Day 0 (N= 65; 66; 65; 63; 74) | 2.7 [2.5 to 2.9] | 2.7 [2.5 to 2.9] | 2.8 [2.5 to 3.1] | 3.1 [2.7 to 3.5] | 2.7 [2.4 to 2.9]
  Month 5 (N= 74; 76; 74; 77; 76) | 55.1 [48.4 to 62.8] | 55.2 [47.9 to 63.6] | 53.7 [46.1 to 62.5] | 49.7 [43.2 to 57.2] | 54.8 [47.3 to 63.5]
  Month 10 (N= 77; 76; 73; 78; 75) | 11.6 [10.0 to 13.6] | 11.6 [9.6 to 14.0] | 9.9 [8.2 to 12.1] | 8.2 [6.8 to 9.8] | 9.8 [8.1 to 11.9]

24. Secondary Outcome: Number of Subjects Seroprotected for Anti-hepatitis B (HBs) Antibodies
Description: Seroprotection is defined as anti-HBs antibody concentration greater than or equal to 10 Milli-International Units per Milliliter (mIU/mL).
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Number; unit: Subjects
Arm/Group | MenHibrix Formulation 1 Group | MenHibrix Formulation 2 Group | MenHibrix Formulation 3 Group | Menjugate Group | ActHIB Group
Number analyzed (Participants) | 74 | 74 | 74 | 76 | 75
Subjects
  Day 0 (N= 57; 55; 56; 52; 57) | 15 | 16 | 12 | 14 | 22
  Month 5 (N= 72; 74; 74; 76; 75) | 71 | 74 | 74 | 76 | 74
  Month 10 (N= 74; 70; 70; 75; 69) | 72 | 68 | 68 | 72 | 68

25. Secondary Outcome: Anti- HBs Antibody Concentrations
Description: Concentrations are presented as GMCs and expressed as Milli-International Units per Milliliter (mIU/mL).
Time Frame: as for outcome 14
Population: as for outcome 19
Measure: Geometric Mean (95% Confidence Interval); unit: Milli-International Units per Milliliter
Arm/Group | MenHibrix Formulation 1 Group | MenHibrix Formulation 2 Group | MenHibrix Formulation 3 Group | Menjugate Group | ActHIB Group
Number analyzed (Participants) | 74 | 74 | 74 | 76 | 75
Milli-International Units per Milliliter
  Day 0 (N= 57; 55; 56; 52; 57) | 13.7 [8.1 to 23.1] | 12.2 [7.8 to 19.2] | 10.0 [6.9 to 14.5] | 10.1 [7.1 to 14.4] | 18.8 [11.1 to 32.0]
  Month 5 (N= 72; 74; 74; 76; 75) | 1769.2 [1276.4 to 2452.2] | 1840.7 [1467.3 to 2309.0] | 1652.6 [1301.2 to 2098.8] | 1752.2 [1373.3 to 2235.6] | 1609.7 [1191.1 to 2175.5]
  Month 10 (N= 74; 70; 70; 75; 69) | 452.3 [311.6 to 656.6] | 490.5 [346.6 to 694.1] | 452.9 [329.7 to 622.3] | 390.5 [278.4 to 547.8] | 534.9 [378.7 to 755.7]

26. Secondary Outcome: Number of Subjects Seroprotected for Anti-poliovirus Types 1, 2 and 3 Antibodies
Description: Seroprotection is defined as anti-polio antibody titer greater than or equal to 1:8 dilution.
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Number; unit: Subjects
Arm/Group | MenHibrix Formulation 1 Group | MenHibrix Formulation 2 Group | MenHibrix Formulation 3 Group | Menjugate Group | ActHIB Group
Number analyzed (Participants) | 71 | 70 | 70 | 76 | 67
Subjects
  Polio-1 Day 0 (N= 56; 58; 50; 56; 52) | 45 | 50 | 44 | 49 | 45
  Polio-1 Month 5 (N= 62; 68; 66; 66; 65) | 62 | 68 | 66 | 66 | 65
  Polio-1 Month 10 (N= 71; 69; 70; 76; 66) | 70 | 65 | 69 | 76 | 65
  Polio-2 Day 0 (N= 56; 59; 50; 55; 52) | 42 | 40 | 36 | 44 | 43
  Polio-2 Month 5 (N= 59; 66; 64; 66; 64) | 59 | 66 | 64 | 66 | 63
  Polio-2 Month 10 (N= 71; 70; 69; 75; 67) | 70 | 66 | 65 | 71 | 64
  Polio-3 Day 0 (N= 56; 59; 50; 56; 52) | 20 | 20 | 24 | 22 | 21
  Polio-3 Month 5 (N= 62; 68; 66; 66; 65) | 62 | 68 | 65 | 65 | 65
  Polio-3 Month 10 (N= 71; 70; 69; 76; 67) | 71 | 69 | 67 | 75 | 65

27. Secondary Outcome: Anti-poliovirus Types 1, 2 and 3 Antibody Titers
Description: Titers are presented as GMTs and expressed in terms of the 50 % inhibitory dilution.
Time Frame: as for outcome 14
Population: as for outcome 19
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | MenHibrix Formulation 1 Group | MenHibrix Formulation 2 Group | MenHibrix Formulation 3 Group | Menjugate Group | ActHIB Group
Number analyzed (Participants) | 71 | 70 | 70 | 76 | 67
Titer
  Polio-1 Day 0 (N= 56; 58; 50; 56; 52) | 36.7 [24.6 to 54.8] | 33.3 [23.2 to 47.6] | 32.9 [21.7 to 49.7] | 52.3 [34.9 to 78.2] | 36.6 [24.6 to 54.3]
  Polio-1 Month 5 (N= 62; 68; 66; 66; 65) | 669.6 [507.5 to 883.4] | 476.8 [364.0 to 624.4] | 574.7 [436.2 to 757.1] | 454.0 [337.5 to 610.7] | 517.6 [396.9 to 674.9]
  Polio-1 Month 10 (N= 71; 69; 70; 76; 66) | 175.8 [129.3 to 239.1] | 120.6 [83.8 to 173.7] | 162.4 [120.2 to 219.4] | 116.4 [86.6 to 156.5] | 166.4 [124.7 to 222.2]
  Polio-2 Day 0 (N= 56; 59; 50; 55; 52) | 14.9 [11.2 to 19.9] | 13.8 [10.3 to 18.3] | 15.9 [11.4 to 22.1] | 17.2 [12.8 to 23.3] | 17.1 [12.7 to 23.0]
  Polio-2 Month 5 (N= 59; 66; 64; 66; 64) | 533.8 [393.3 to 724.4] | 369.8 [273.4 to 500.0] | 408.0 [297.6 to 559.4] | 348.9 [265.3 to 458.8] | 368.0 [264.0 to 512.9]
  Polio-2 Month 10 (N= 71; 70; 69; 75; 67) | 139.8 [104.1 to 187.8] | 94.1 [67.5 to 131.3] | 110.1 [77.0 to 157.4] | 89.6 [63.4 to 126.7] | 88.3 [61.6 to 126.5]
  Polio-3 Day 0 (N= 56; 59; 50; 56; 52) | 6.4 [5.3 to 7.8] | 6.6 [5.2 to 8.3] | 7.9 [6.2 to 10.1] | 7.7 [5.8 to 10.1] | 8.0 [6.1 to 10.5]
  Polio-3 Month 5 (N= 62; 68; 66; 66; 65) | 1266.3 [992.1 to 1616.2] | 1034.8 [778.8 to 1374.8] | 1062.2 [809.2 to 1394.2] | 1084.9 [804.2 to 1463.7] | 945.5 [695.9 to 1284.5]
  Polio-3 Month 10 (N= 71; 70; 69; 76; 67) | 348.4 [260.0 to 466.9] | 263.8 [194.2 to 358.3] | 250.9 [184.1 to 342.1] | 264.0 [192.1 to 362.9] | 203.9 [139.6 to 297.8]

28. Secondary Outcome: Number of Subjects With Anti-pneumococcal Antibody Concentrations Greater Than or Equal to Pre-defined Cut-off Values
Description: Pneumococcal antibodies assessed included anti-4, anti-6B, anti-9V, anti-14, anti-18C, anti-19F and anti-23F antibodies. The cut-off values assessed were 0.05 and 0.2 micrograms per milliliter (µg/mL).
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Number; unit: Subjects
Arm/Group | MenHibrix Formulation 1 Group | MenHibrix Formulation 2 Group | MenHibrix Formulation 3 Group | Menjugate Group | ActHIB Group
Number analyzed (Participants) | 73 | 71 | 72 | 77 | 67
Subjects
  Anti-4 ≥ 0.05 µg/mL Day 0 (N=44;43;39;51;46) | 10 | 9 | 10 | 11 | 10
  Anti-4 ≥ 0.05 µg/mL Month 5 (N=69;70;69;58;66) | 69 | 70 | 69 | 2 | 66
  Anti-4 ≥ 0.05 µg/mL Month 10 (N=70;68;66;69;64) | 70 | 68 | 65 | 1 | 64
  Anti-6B ≥ 0.05 µg/mL Day 0 (N=44;41;39;49;49) | 18 | 21 | 20 | 25 | 23
  Anti-6B ≥ 0.05 µg/mL Month 5 (N=68;70;69;63;65) | 65 | 69 | 61 | 3 | 60
  Anti-6B ≥ 0.05 µg/mL Month 10 (N=69;63;62;71;62) | 62 | 57 | 55 | 2 | 55
  Anti-9V ≥ 0.05 µg/mL Day 0 (N=46;42;40;52;48) | 19 | 22 | 23 | 23 | 18
  Anti-9V ≥ 0.05 µg/mL Month 5 (N=68;71;71;62;67) | 68 | 70 | 71 | 3 | 66
  Anti-9V ≥ 0.05 µg/mL Month 10 (N=60;60;56;63;56) | 60 | 58 | 56 | 5 | 56
  Anti-14 ≥ 0.05 µg/mL Day 0 (N=31;33;31;41;43) | 29 | 25 | 26 | 37 | 39
  Anti-14 ≥ 0.05 µg/mL Month 5 (N=65;65;68;49;65) | 65 | 65 | 68 | 24 | 65
  Anti-14 ≥ 0.05 µg/mL Month 10 (N=68;67;64;69;61) | 67 | 67 | 63 | 13 | 61
  Anti-18C ≥ 0.05 µg/mL Day 0 (N=40;40;37;47;47) | 20 | 19 | 21 | 23 | 25
  Anti-18C ≥ 0.05 µg/mL Month 5 (N=67;71;72;65;67) | 66 | 71 | 72 | 5 | 66
  Anti-18C ≥ 0.05 µg/mL Month 10 (N=48;52;51;53;46) | 47 | 52 | 51 | 0 | 45
  Anti-19F ≥ 0.05 µg/mL Day 0 (N=42;42;36;50;45)) | 28 | 28 | 25 | 37 | 28
  Anti-19F ≥ 0.05 µg/mL Month 5 (N=65;67;66;56;65) | 65 | 66 | 66 | 7 | 65
  Anti-19F ≥ 0.05 µg/mL Month 10 (N=73;71;65;77;63) | 73 | 68 | 65 | 14 | 61
  Anti-23F ≥ 0.05 µg/mL Day 0 (N=41;43;38;48;48) | 17 | 14 | 15 | 19 | 22
  Anti-23F ≥ 0.05 µg/mL Month 5 (N=66;68;70;59;66) | 65 | 66 | 67 | 3 | 63
  Anti-23F ≥ 0.05 µg/mL Month 10 (N=73;69;63;75;65) | 71 | 67 | 59 | 0 | 63
  Anti-4 ≥ 0.2 µg/mL Day 0 (N=44;43;39;51;46) | 3 | 1 | 3 | 1 | 2
  Anti-4 ≥ 0.2 µg/mL Month 5 (N=69;70;69;58;66) | 69 | 70 | 69 | 1 | 66
  Anti-4 ≥ 0.2 µg/mL Month 10 (N=70;68;66;69;64) | 65 | 60 | 61 | 1 | 53
  Anti-6B ≥ 0.2 µg/mL Day 0 (N=44;41;39;49;49) | 6 | 11 | 7 | 9 | 8
  Anti-6B ≥ 0.2 µg/mL Month 5 (N=68;70;69;63;65) | 58 | 64 | 56 | 1 | 56
  Anti-6B ≥ 0.2 µg/mL Month 10 (N=69;63;62;71;62) | 45 | 41 | 49 | 0 | 42
  Anti-9V ≥ 0.2 µg/mL Day 0 (N=46;42;40;52;48) | 9 | 6 | 8 | 10 | 8
  Anti-9V ≥ 0.2 µg/mL Month 5 (N=68;71;71;62;67) | 68 | 69 | 71 | 1 | 66
  Anti-9V ≥ 0.2 µg/mL Month 10 (N=60;60;56;63;56) | 55 | 54 | 55 | 2 | 56
  Anti-14 ≥ 0.2 µg/mL Day 0 (N=31;33;31;41;43) | 20 | 18 | 16 | 28 | 30
  Anti-14 ≥ 0.2 µg/mL Month 5 (N=65;65;68;49;65) | 64 | 65 | 68 | 7 | 64
  Anti-14 ≥ 0.2 µg/mL Month 10 (N=68;67;64;69;61) | 64 | 65 | 63 | 5 | 60
  Anti-18C ≥ 0.2 µg/mL Day 0 (N=40;40;37;47;47) | 10 | 6 | 8 | 6 | 10
  Anti-18C ≥ 0.2 µg/mL Month 5 (N=67;71;72;65;67) | 66 | 70 | 72 | 2 | 65
  Anti-18C ≥ 0.2 µg/mL Month 10 (N=48;52;51;53;46) | 47 | 50 | 50 | 0 | 42
  Anti-19F ≥ 0.2 µg/mL Day 0 (N=42;42;36;50;45) | 14 | 18 | 16 | 22 | 15
  Anti-19F ≥ 0.2 µg/mL Month 5 (N=65;67;66;56;65) | 65 | 66 | 66 | 2 | 63
  Anti-19F ≥ 0.2 µg/mL Month 10 (N=73;71;65;77;63) | 54 | 51 | 55 | 8 | 45
  Anti-23F ≥ 0.2 µg/mL Day 0 (N=41;43;38;48;48) | 5 | 6 | 7 | 9 | 8
  Anti-23F ≥ 0.2 µg/mL Month 5 (N=66;68;70;59;66) | 64 | 64 | 67 | 0 | 62
  Anti-23F ≥ 0.2 µg/mL Month 10 (N=73;69;63;75;65) | 66 | 56 | 53 | 0 | 52

29. Secondary Outcome: Anti-pneumococcal Antibody Concentrations
Description: Pneumococcal antibodies assessed included anti-4, anti-6B, anti-9V, anti-14, anti-18C, anti-19F and anti-23F antibodies. Concentrations are presented as GMCs and expressed as micrograms per milliliter (µg/mL).
Time Frame: as for outcome 14
Population: as for outcome 19
Measure: Geometric Mean (95% Confidence Interval); unit: Micrograms per milliliter (µg/mL)
Arm/Group | MenHibrix Formulation 1 Group | MenHibrix Formulation 2 Group | MenHibrix Formulation 3 Group | Menjugate Group | ActHIB Group
Number analyzed (Participants) | 73 | 71 | 72 | 77 | 67
Micrograms per milliliter (µg/mL)
  Anti-4 Day 0 (N= 44; 43; 39; 51; 46) | 0.036 [0.029 to 0.046] | 0.035 [0.028 to 0.043] | 0.040 [0.030 to 0.053] | 0.034 [0.028 to 0.040] | 0.036 [0.029 to 0.046]
  Anti-4 Month 5 (N= 69; 70; 69; 58; 66) | 2.101 [1.780 to 2.480] | 2.049 [1.718 to 2.442] | 2.023 [1.729 to 2.366] | 0.027 [0.024 to 0.030] | 2.062 [1.787 to 2.380]
  Anti-4 Month 10 (N= 70; 68; 66; 69; 64) | 0.495 [0.407 to 0.603] | 0.528 [0.431 to 0.646] | 0.508 [0.414 to 0.623] | 0.026 [0.024 to 0.027] | 0.450 [0.372 to 0.544]
  Anti-6B Day 0 (N= 44; 41; 39; 49; 49) | 0.055 [0.039 to 0.078] | 0.080 [0.052 to 0.123] | 0.067 [0.046 to 0.099] | 0.070 [0.049 to 0.101] | 0.067 [0.045 to 0.099]
  Anti-6B Month 5 (N= 68; 70; 69; 63; 65) | 1.060 [0.744 to 1.511] | 1.079 [0.808 to 1.442] | 0.834 [0.567 to 1.225] | 0.027 [0.025 to 0.030] | 0.879 [0.604 to 1.278]
  Anti-6B Month 10 (N= 69; 63; 62; 71; 62) | 0.307 [0.223 to 0.424] | 0.307 [0.223 to 0.423] | 0.292 [0.215 to 0.398] | 0.026 [0.025 to 0.027] | 0.308 [0.220 to 0.430]
  Anti-9V Day 0 (N= 46; 42; 40; 52; 48) | 0.058 [0.040 to 0.085] | 0.065 [0.044 to 0.096] | 0.079 [0.051 to 0.121] | 0.059 [0.043 to 0.080] | 0.055 [0.039 to 0.077]
  Anti-9V Month 5 (N= 68; 71; 71; 62; 67) | 3.102 [2.563 to 3.754] | 2.363 [1.822 to 3.066] | 2.823 [2.376 to 3.354] | 0.028 [0.024 to 0.033] | 2.651 [2.079 to 3.380]
  Anti-9V Month 10 (N= 60; 60; 56; 63; 56) | 0.818 [0.656 to 1.020] | 0.721 [0.555 to 0.937] | 0.933 [0.758 to 1.147] | 0.030 [0.025 to 0.035] | 0.881 [0.742 to 1.045]
  Anti-14 Day 0 (N= 31; 33; 31; 41; 43) | 0.367 [0.203 to 0.664] | 0.227 [0.121 to 0.427] | 0.258 [0.143 to 0.467] | 0.394 [0.253 to 0.612] | 0.388 [0.247 to 0.609]
  Anti-14 Month 5 (N= 65; 65; 68; 49; 65) | 4.095 [3.037 to 5.520] | 5.592 [4.238 to 7.378] | 4.309 [3.306 to 5.616] | 0.062 [0.043 to 0.090] | 4.372 [3.211 to 5.954]
  Anti-14 Month 10 (N= 68; 67; 64; 69; 61) | 2.362 [1.786 to 3.124] | 2.767 [2.149 to 3.563] | 2.549 [1.968 to 3.304] | 0.039 [0.030 to 0.051] | 2.379 [1.807 to 3.132]
  Anti-18C Day 0 (N= 40; 40; 37; 47; 47) | 0.073 [0.049 to 0.109] | 0.063 [0.045 to 0.090] | 0.075 [0.050 to 0.111] | 0.063 [0.045 to 0.090] | 0.078 [0.054 to 0.112]
  Anti-18C Month 5 (N= 67; 71; 72; 65; 67) | 3.518 [2.748 to 4.504] | 2.969 [2.464 to 3.578] | 2.936 [2.440 to 3.533] | 0.029 [0.025 to 0.035] | 3.326 [2.557 to 4.327]
  Anti-18C Month 10 (N= 48; 52; 51; 53; 46) | 0.775 [0.601 to 1.000] | 0.742 [0.607 to 0.907] | 0.708 [0.577 to 0.867] | 0.025 [0.025 to 0.025] | 0.668 [0.503 to 0.887]
  Anti-19F Day 0 (N= 42; 42; 36; 50; 45) | 0.124 [0.076 to 0.202] | 0.126 [0.083 to 0.190] | 0.129 [0.080 to 0.206] | 0.135 [0.092 to 0.198] | 0.115 [0.073 to 0.180]
  Anti-19F Month 5 (N= 65; 67; 66; 56; 65) | 2.303 [1.889 to 2.806] | 1.846 [1.444 to 2.360] | 2.061 [1.719 to 2.472] | 0.030 [0.026 to 0.035] | 1.881 [1.508 to 2.346]
  Anti-19F Month 10 (N= 73; 71; 65; 77; 63) | 0.413 [0.320 to 0.532] | 0.335 [0.252 to 0.443] | 0.397 [0.307 to 0.512] | 0.042 [0.031 to 0.056] | 0.339 [0.252 to 0.456]
  Anti-23F Day 0 (N= 41; 43; 38; 48; 48) | 0.053 [0.038 to 0.075] | 0.045 [0.033 to 0.062] | 0.062 [0.040 to 0.096] | 0.060 [0.041 to 0.086] | 0.065 [0.044 to 0.098]
  Anti-23F Month 5 (N= 66; 68; 70; 59; 66) | 2.581 [1.970 to 3.381] | 2.112 [1.544 to 2.891] | 2.098 [1.551 to 2.838] | 0.027 [0.025 to 0.029] | 1.988 [1.426 to 2.772]
  Anti-23F Month 10 (N= 73; 69; 63; 75; 65) | 0.783 [0.595 to 1.032] | 0.642 [0.474 to 0.870] | 0.644 [0.469 to 0.885] | 0.025 [0.025 to 0.025] | 0.578 [0.426 to 0.785]

30. Secondary Outcome: Number of Subjects Reporting Solicited Local and General Symptoms During the Primary Vaccination Course
Description: Solicited local symptoms assessed include pain, redness and swelling at the injection site. Solicited general symptoms assessed include drowsiness, irritability, loss of appetite and fever (rectal temperature greater than or equal to 38 degrees Celcius).
Time Frame: During the 8-Day (Day 0-7) follow-up period after any vaccine dose during the primary vaccination course
Population: The analysis was performed on the Total Vaccinated Cohort, on subjects having completed the symptom sheet.
Measure: Number; unit: Subjects
Arm/Group | MenHibrix Formulation 1 Group | MenHibrix Formulation 2 Group | MenHibrix Formulation 3 Group | Menjugate Group | ActHIB Group
Number analyzed (Participants) | 81 | 82 | 79 | 81 | 82
Subjects
  Pain | 54 | 50 | 53 | 66 | 60
  Redness | 67 | 67 | 64 | 75 | 69
  Swelling | 53 | 64 | 56 | 60 | 58
  Drowsiness | 65 | 72 | 58 | 70 | 67
  Irritability | 76 | 79 | 76 | 80 | 80
  Loss of appetite | 57 | 56 | 49 | 47 | 58
  Fever | 65 | 64 | 64 | 64 | 70

31. Secondary Outcome: Number of Subjects Reporting Solicited Local and General Symptoms After Administration of the Polysaccharide Challenge Dose
Description: as for outcome 30
Time Frame: During the 8-Day (Day 0-7) follow-up period after the polysaccharide challenge dose
Population: The analysis was performed on the Booster Total Vaccinated Cohort, on subjects having completed the symptom sheet.
Measure: Number; unit: Subjects
Arm/Group | MenHibrix Formulation 1 Group | MenHibrix Formulation 2 Group | MenHibrix Formulation 3 Group | Menjugate Group | ActHIB Group
Number analyzed (Participants) | 80 | 79 | 77 | 81 | 77
Subjects
  Pain | 19 | 15 | 18 | 17 | 16
  Redness | 39 | 27 | 27 | 44 | 29
  Swelling | 15 | 15 | 13 | 15 | 12
  Drowsiness | 26 | 25 | 17 | 26 | 18
  Irritability | 48 | 48 | 45 | 46 | 49
  Loss of appetite | 26 | 27 | 25 | 24 | 23
  Fever | 29 | 20 | 27 | 36 | 34

32. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events During the Primary Vaccination Course
Description: Unsolicited adverse event covers any adverse event reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: During the 31-Day (Day 0-30) follow-up period after any vaccine dose during the primary vaccination course
Population: The analysis was performed on the Total Vaccinated Cohort.
Measure: Number; unit: Subjects
Arm/Group | MenHibrix Formulation 1 Group | MenHibrix Formulation 2 Group | MenHibrix Formulation 3 Group | Menjugate Group | ActHIB Group
Number analyzed (Participants) | 82 | 82 | 80 | 81 | 82
Subjects | 64 | 68 | 56 | 58 | 68

33. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events After Administration of the Polysaccharide Challenge Dose
Description: as for outcome 32
Time Frame: During the 31-Day (Day 0-30) follow-up period after administration of the polysaccharide challenge dose
Population: The analysis was performed on the Booster Total Vaccinated Cohort.
Measure: Number; unit: Subjects
Arm/Group | MenHibrix Formulation 1 Group | MenHibrix Formulation 2 Group | MenHibrix Formulation 3 Group | Menjugate Group | ActHIB Group
Number analyzed (Participants) | 80 | 79 | 77 | 81 | 77
Subjects | 39 | 46 | 47 | 50 | 52

34. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events During the Primary Vaccination Course
Description: Serious adverse events cover all medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: Up to one month after the 3-dose primary vaccination course (Month 5)
Population: The analysis was performed on the Total Vaccinated Cohort.
Measure: Number; unit: Subjects
Arm/Group | MenHibrix Formulation 1 Group | MenHibrix Formulation 2 Group | MenHibrix Formulation 3 Group | Menjugate Group | ActHIB Group
Number analyzed (Participants) | 82 | 82 | 80 | 81 | 82
Subjects | 5 | 5 | 2 | 4 | 6

35. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events After Administration of the Polysaccharide Challenge Dose
Description: as for outcome 34
Time Frame: Up to one month following administration of the polysaccharide challenge dose (Month 11)
Population: The analysis was performed on the Booster Total Vaccinated Cohort.
Measure: Number; unit: Subjects
Arm/Group | MenHibrix Formulation 1 Group | MenHibrix Formulation 2 Group | MenHibrix Formulation 3 Group | Menjugate Group | ActHIB Group
Number analyzed (Participants) | 80 | 79 | 77 | 81 | 77
Subjects | 0 | 0 | 0 | 0 | 2

ADVERSE EVENTS:
Time Frame: SAEs: Up to 1 month following primary vaccination and challenge dose; Non-systematically assessed other AEs: Up to 31 days following primary vaccination and challenge dose; Systematically assessed other AEs: During 8-day follow-up after each dose.
Description: The number at risk for systematically assessed symptoms comprises only those subjects who had returned the symptom sheet.
Arm/Group | MenHibrix Formulation 1 Group | MenHibrix Formulation 2 Group | MenHibrix Formulation 3 Group | Menjugate Group | ActHIB Group
Serious Adverse Events (participants affected / at risk) | 5/82 | 5/82 | 2/80 | 4/81 | 6/82
Other Adverse Events (participants affected / at risk) | 81/82 | 81/82 | 77/80 | 81/81 | 82/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | MenHibrix Formulation 1 Group (N=82) | MenHibrix Formulation 2 Group (N=82) | MenHibrix Formulation 3 Group (N=80) | Menjugate Group (N=81) | ActHIB Group (N=82)
Balanitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 — Following primary vaccination
Bronchiolitis (Infections and infestations) | 1 | 1 | 1 | 0 | 4 — Following primary vaccination
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 — Following primary vaccination
Croup infectious (Infections and infestations) | 0 | 1 | 0 | 0 | 0 — Following primary vaccination
Deafness (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 — Following primary vaccination
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 — Following primary vaccination
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 — Following primary vaccination
Gastroenteritis viral (Infections and infestations) | 2 | 0 | 0 | 1 | 0 — Following primary vaccination
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 — Following primary vaccination
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0 — Following primary vaccination
Lobar pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 — Following primary vaccination
Milk allergy (Immune system disorders) | 0 | 1 | 0 | 0 | 0 — Following primary vaccination
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 1 | 0 — Following primary vaccination
Sudden infant death syndrome (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 — Following primary vaccination
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 — Following primary vaccination
Bronchiolitis (Infections and infestations) | 0/80 | 0/79 | 0/77 | 0 | 1/77 — Following challenge dose administration
Pneumonia (Infections and infestations) | 0/80 | 0/79 | 0/77 | 0 | 1/77 — Following challenge dose administration
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | MenHibrix Formulation 1 Group (N=82) | MenHibrix Formulation 2 Group (N=82) | MenHibrix Formulation 3 Group (N=80) | Menjugate Group (N=81) | ActHIB Group (N=82)
Upper respiratory tract infection (Infections and infestations) | 19 | 24 | 24 | 25 | 31 — Following primary vaccination
Injection site bruising (General disorders) | 12 | 12 | 15 | 16 | 11 — Following primary vaccination
Irritability (Psychiatric disorders) | 13 | 6 | 9 | 5 | 12 — Following primary vaccination
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 | 9 | 4 | 10 | 6 — Following primary vaccination
Vomiting (Gastrointestinal disorders) | 6 | 9 | 7 | 3 | 9 — Following primary vaccination
Diarrhoea (Gastrointestinal disorders) | 6 | 10 | 6 | 7 | 4 — Following primary vaccination
Pyrexia (General disorders) | 7 | 8 | 3 | 2 | 8 — Following primary vaccination
Teething (Gastrointestinal disorders) | 7 | 6 | 3 | 2 | 7 — Following primary vaccination
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 4 | 5 | 4 — Following primary vaccination
Rash (Skin and subcutaneous tissue disorders) | 8 | 2 | 7 | 3 | 2 — Following primary vaccination
Gingival pain (Gastrointestinal disorders) | 1 | 3 | 3 | 5 | 2 — Following primary vaccination
Bronchiolitis (Infections and infestations) | 3 | 4 | 3 | 0 | 5 — Following primary vaccination
Rhinitis (Infections and infestations) | 0 | 3 | 4 | 3 | 0 — Following primary vaccination
Eczema (Skin and subcutaneous tissue disorders) | 4 | 6 | 2 | 0 | 4 — Following primary vaccination
Upper respiratory tract infection (Infections and infestations) | 12/80 | 10/79 | 14/77 | 17 | 11/77 — Following challenge dose administration
Injection site haemorrhage (General disorders) | 7/80 | 9/79 | 3/77 | 7 | 7/77 — Following challenge dose administration
Irritability (Psychiatric disorders) | 5/80 | 6/79 | 8/77 | 6 | 6/77 — Following challenge dose administration
Rhinorhea (Respiratory, thoracic and mediastinal disorders) | 4/80 | 6/79 | 5/77 | 7 | 5/77 — Following challenge dose administration
Pyrexia (General disorders) | 2/80 | 4/79 | 10/77 | 3 | 6/77 — Following challenge dose administration
Teething (Gastrointestinal disorders) | 2/80 | 5/79 | 4/77 | 6 | 7/77 — Following challenge dose administration
Vomiting (Gastrointestinal disorders) | 4/80 | 4/79 | 3/77 | 3 | 5/77 — Following challenge dose administration
Cough (Respiratory, thoracic and mediastinal disorders) | 2/80 | 6/79 | 3/77 | 3 | 3/77 — Following challenge dose administration
Otitis media (Infections and infestations) | 5/80 | 3/79 | 3/77 | 1 | 3/77 — Following challenge dose administration
Diarrhea (Gastrointestinal disorders) | 4/80 | 0/79 | 2/77 | 5 | 0/77 — Following challenge dose administration
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0/80 | 1/79 | 4/77 | 0 | 0/77 — Following challenge dose administration
Insomnia (Psychiatric disorders) | 0/80 | 1/79 | 1/77 | 1 | 4/77 — Following challenge dose administration
Pain at the injection site (General disorders) | 54/81 | 50 | 53/79 | 66 | 60 — Following primary vaccination
Redness at the injection site (General disorders) | 67/81 | 67 | 64/79 | 75 | 69 — Following primary vaccination
Swelling at the injection site (General disorders) | 53/81 | 64 | 56/79 | 60 | 58 — Following primary vaccination
Drowsiness (General disorders) | 65/81 | 72 | 58/78 | 70 | 67 — Following primary vaccination
Irritability (General disorders) | 76/81 | 79 | 76/78 | 80 | 80 — Following primary vaccination
Loss of appetite (General disorders) | 57/81 | 56 | 49/78 | 47 | 58 — Following primary vaccination
Fever (General disorders) | 65/81 | 64 | 64/78 | 64 | 70 — Following primary vaccination
Pain at the injection site (General disorders) | 19/80 | 15/79 | 18/77 | 17 | 16/77 — Following challenge dose administration
Redness at the injection site (General disorders) | 39/80 | 27/79 | 27/77 | 44 | 29/77 — Following challenge dose administration
Swelling at the injection site (General disorders) | 15/80 | 15/79 | 13/77 | 15 | 12/77 — Following challenge dose administration
Drowsiness (General disorders) | 26/80 | 25/79 | 17/77 | 26 | 18/77 — Following challenge dose administration
Irritability (General disorders) | 48/80 | 48/79 | 45/77 | 46 | 49/77 — Following challenge dose administration
Loss of appetite (General disorders) | 26/80 | 27/79 | 25/77 | 24 | 23/77 — Following challenge dose administration
Fever (General disorders) | 29/80 | 20/79 | 27/77 | 36 | 34/77 — Following challenge dose administration

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.